CLINICAL TRIAL: NCT01514253
Title: Reduced Infant Response to a Routine Care Procedure After Glucose 25% Analgesia in Comparison to Materna RTF Stage 1
Acronym: glucose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Shay Barak, Senior Neonatologist, Neonatal Intensive Care, The Baruch Padeh Medical Center, Poriya
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SAOR 006.CTIL
Record Dates: First submitted 2012-01-05; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Infant, Newborn, Diseases
Keywords: glucose; analgesic; newborns
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- glucose 25% (Experimental): 1 ml of glucose once
  Interventions: Drug: Glucose 25%
- infant formula (Experimental): Materna RTF stage 1
  Interventions: Dietary Supplement: Materna RTF Stage 1
- Water for Injection (Placebo Comparator): 1 ml Water for Injection (WFI), 2-3 minutes prior red-reflex examination
  Interventions: Other: Water for Injection

INTERVENTIONS:
Drug: Glucose 25% — 1 ml glucose 25%, once
  Arms: glucose 25%
Dietary Supplement: Materna RTF Stage 1 — 1ml Materna RTF Phase 1, 2-3 minutes prior red-reflex examination.
  Other Names: Materna RTF Phase 1
  Arms: infant formula
Other: Water for Injection — 1 ml Water for Injection (WFI), 2-3 minutes prior red-reflex examination
  Other Names: WFI
  Arms: Water for Injection

SUMMARY:
Glucose has analgesic and calming effects in newborns. To date, it is not known whether the beneficial effects extend to care giving procedures that are performed after painful procedures. The investigators objective is to determine the effect of glucose 25% analgesia in comparison to Materna RTF Stage 1 for procedural pain on infant pain responses during a subsequent care giving procedure.

DETAILED DESCRIPTION:
During hospitalization, a neonate undergoes a number of necessary procedures that may be either painful or cause discomfort to the baby.

Pain experienced during the neonatal period is known to have long term effects on the baby.

The red-reflex test is a routine examination performed on a neonate after birth and once again before discharge from the hospital. The examination causes discomfort to the infant Glucose has analgesic and calming effects in newborns. To date, it is not known whether the beneficial effects extend to care giving procedures that are performed after painful procedures. The investigators objective is to determine the effect of glucose 25% analgesia in comparison to Materna RTF Stage 1 for procedural pain on infant pain responses during a subsequent care giving procedure.

ELIGIBILITY:
Inclusion Criteria:

* Full term above 37 weeks gestation.
* Normal birth-weight, healthy infants
* Males and Females
* Whose parents have signed the informed consent form

Exclusion Criteria:

* Premature born below 37 weeks
* Chromosomal abnormalities or congenital malformation.
* Suffering neurological imbalance
* Inability of oral feeding

Ages: 1 Day to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
less discomfort | immediate, during examination (day 1)
  the infant will experience less pain during examination

CONTACTS AND LOCATIONS:
Overall Officials: Shay Barak, MD, Principal Investigator — The Baruch Pade Medical Center - Poriya; Amir Kushnir, MD, Study Director — The Baruch Padeh Medical Center - Poria
Locations (1):
- NICU Department, The Baruch Padeh medical Center - Poriya, Tiberias, Israel